CLINICAL TRIAL: NCT01693692
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study of TD-9855 in Patients With Fibromyalgia (FM)
Brief Title: Phase 2 Study of TD-9855 to Treat Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0092
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TD-9855 Group 1 (Experimental): Group 1 to be dosed with TD-9855
  Interventions: Drug: TD-9855 Group 1
- TD-9855 Group 2 (Experimental): Group 2 to be dosed with TD-9855
  Interventions: Drug: TD-9855 Group 2
- Placebo (Placebo Comparator): Group to be dosed with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-9855 Group 1
  Arms: TD-9855 Group 1
Drug: TD-9855 Group 2
  Arms: TD-9855 Group 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study study is to determine whether TD-9855 is effective in treating patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* • American College of Rheumatology (ACR) Diagnostic Criteria for Fibromyalgia (FM)

  * Informed consent
  * 18 to 65 years of age
  * Discontinue therapy with adrenergic-acting drugs, and certain other medications

    * Only acetaminophen or NSAID as rescue pain medication
    * No narcotic pain meds or benzodiazepines
    * Only non-benzodiazepines as rescue hypnotics

Exclusion Criteria:

* Any current psychiatric disorder, lifetime bipolar disorder, severe comorbid Axis II disorder, mental retardation, etc, as assessed by Mini International Neuropsychiatric Interview (MINI)
* Major depression at screening by MINI when unable to be washed out of MDD meds (investigator or provider's judgment)
* Risk of suicide (investigator opinion and/or C-SSRS)
* Recent history of substance or alcohol abuse
* BMI <18 or ≥45
* Concurrent disease; pain for diagnosed illness other than FM; non-compliance; history of seizures; pheochromocytoma; glaucoma; CV disease; orthostatic hypotension or orthostatic tachycardia; untreated sleep apnea
* Abnormal lab values (liver, kidney, thyroid, and others)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (34):
- United States (34):
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - TriWest Research Associates, LLC, El Cajon, California
  - Arroyo Medical Group, Inc., Pismo Beach, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Meridien Research, Lakeland, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - GTC Research, Shawnee Mission, Kansas
  - Beacon Clinical Research, Brockton, Massachusetts
  - Beacon Clinical Research, New Bedford, Massachusetts
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Wake Research Associates, Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Clinical Research Source, Inc., Perrysburg, Ohio
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Carolina Center for Rheumatology & Arthritis Care, Rock Hill, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Swedish Rheumatology Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

REFERENCES:
- [Derived] Kanodia J, Lo A, Baldwin RM, Graham RA, Bourdet DL. Pharmacokinetics of Ampreloxetine, a Norepinephrine Reuptake Inhibitor, in Healthy Subjects and Adults with Attention-Deficit/Hyperactive Disorder or Fibromyalgia Pain. Clin Pharmacokinet. 2021 Jan;60(1):121-131. doi: 10.1007/s40262-020-00918-7. PMID 32856281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 392 participants were enrolled across 53 study sites in the United States.
Pre-assignment Details: 392 participants were enrolled, but 9 participants were not treated with the study drug.
Groups:
- Placebo: Participants will be administered a placebo once daily for 6 weeks.
- TD-9855 Group 1: Participants will be administered TD-9855 at an initial dose of 2.5 mg once daily for 1 week, before increasing the dose to 5 mg once daily for the following 5 weeks. Participants who are unable to tolerate the initial dose level will be discontinued from further dosing and will be considered to have withdrawn prematurely from the study.
- TD-9855 Group 2: Participants will be administered TD-9855 at an initial dose of 10 mg once daily for 1 week, before increasing the dose to 20 mg once daily for the following 5 weeks. Participants who are unable to tolerate the initial dose level will be discontinued from further dosing and will be considered to have withdrawn prematurely from the study.
Period: Overall Study
Arm/Group | Placebo | TD-9855 Group 1 | TD-9855 Group 2
Started | 130 | 131 | 131
Received Study Drug | 128 | 127 | 128
Completed | 100 | 97 | 95
Not Completed | 30 | 34 | 36
Not completed — Withdrawal by Subject | 12 | 10 | 11
Not completed — Adverse Event | 7 | 14 | 9
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 5 | 4 | 6
Not completed — Lost to Follow-up | 2 | 2 | 3
Not completed — Other | 4 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TD-9855 Group 1 | TD-9855 Group 2 | Total
Number analyzed (Participants) | 130 | 131 | 131 | 392
Age, Continuous [Mean (Full Range); unit: years] | 45.8 [18.0 to 65.0] | 48.0 [19.0 to 65.0] | 43.2 [19.0 to 65.0] | 45.7 [18.0 to 65.0]
Age, Customized [Count of Participants; unit: Participants]
  Age (years): 18 - 45 Years of Age | 55 | 51 | 73 | 179
  Age (years): 46 - 65 Years of Age | 75 | 80 | 58 | 213
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 123 | 123 | 369
  Male | 7 | 8 | 8 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 16 | 19 | 57
  Not Hispanic or Latino | 106 | 115 | 112 | 333
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 13 | 18 | 20 | 51
  White | 110 | 107 | 107 | 324
  More than one race | 2 | 6 | 1 | 9
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 130 | 131 | 131 | 392
Weight [Mean (Standard Deviation); unit: kg] | 81.9 (17.64) | 83.2 (17.68) | 79.0 (17.27) | 81.4 (17.57)
Height [Mean (Standard Deviation); unit: cm] | 163.3 (6.85) | 164.5 (7.65) | 164.0 (8.49) | 164.0 (7.69)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (6.24) | 30.7 (5.74) | 29.3 (5.59) | 30.2 (5.89)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Pain Score Based on the Mean of the Last 7 Daily Pain Numeric Rating Scale (NRS) Scores From the Daily Pain Diaries
Description: Pain NRS score is based on an 11-point scale where 0 represents no pain and 10 represents the worst possible pain.
Time Frame: Baseline and Week 6
Population: Only participants with available data were used for this analysis.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | TD-9855 Group 1 | TD-9855 Group 2
Number analyzed (Participants) | 126 | 122 | 125
percentage change | -0.9 (0.17) | -1.2 (0.18) | -1.4 (0.17)
Statistical Analysis 1: Comparison: Placebo vs TD-9855 Group 1; Test type: Superiority; p = 0.1683, ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 1-sided [upper limit 0.2], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Placebo vs TD-9855 Group 2; Test type: Superiority; p = 0.0277, ANCOVA; Mean Difference (Final Values) = -0.47, 95% CI 1-sided [upper limit -0.1], Standard Error of Mean 0.25

2. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQ)
Description: FIQ score is based on the total score from 0 to 100 gained from 10 questions, where a lower total score represents less impact from fibromyalgia.
Time Frame: Day 43 (End of study treatment)
Population: Only participants with available data were used for this analysis.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TD-9855 Group 1 | TD-9855 Group 2
Number analyzed (Participants) | 126 | 122 | 125
score on a scale | 44.0 (1.75) | 42.4 (1.75) | 38.2 (1.75)
Statistical Analysis 1: Comparison: Placebo vs TD-9855 Group 1; Test type: Superiority; p = 0.2637, ANCOVA; Mean Difference (Final Values) = -1.57, 95% CI 1-sided [upper limit 2.5], Standard Error of Mean 2.48
Statistical Analysis 2: Comparison: Placebo vs TD-9855 Group 2; Test type: Superiority; p = 0.0097, ANCOVA; Mean Difference (Final Values) = -5.80, 95% CI 1-sided [upper limit -1.7], Standard Error of Mean 2.47

3. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: PGIC score is based on a 7-category scale where a score of 1 indicates the participant's condition is very much improved, and a score of 7 indicates the participant's condition is very much worse.
Time Frame: Day 43 (End of study treatment)
Population: Only participants with available data were used for this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TD-9855 Group 1 | TD-9855 Group 2
Number analyzed (Participants) | 126 | 122 | 125
score on a scale | 3.2 (0.11) | 2.9 (0.11) | 2.8 (0.11)
Statistical Analysis 1: Comparison: Placebo vs TD-9855 Group 1; Test type: Superiority; p = 0.0639, ANCOVA; Mean Difference (Final Values) = -0.24, 95% CI 1-sided [upper limit 0.0], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs TD-9855 Group 2; Test type: Superiority; p = 0.0070, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI 1-sided [upper limit -0.1], Standard Error of Mean 0.16

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 63
Description: Only data from participants who received study drug or placebo is included here.
Arm/Group | Placebo | TD-9855 Group 1 | TD-9855 Group 2
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/127 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/128 | 1/127 | 1/128
Other Adverse Events (participants affected / at risk) | 71/128 | 78/127 | 90/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | TD-9855 Group 1 (N=127) | TD-9855 Group 2 (N=128)
Transient neurological symptoms of unknown etiology (Nervous system disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | TD-9855 Group 1 (N=127) | TD-9855 Group 2 (N=128)
Headache (Nervous system disorders) | 10 | 10 | 17
Nausea (Gastrointestinal disorders) | 9 | 11 | 10
Dizziness (Nervous system disorders) | 5 | 7 | 13
Insomnia (General disorders) | 4 | 7 | 11
Constipation (Gastrointestinal disorders) | 1 | 6 | 12
Fatigue (General disorders) | 4 | 6 | 9
Urinary tract infection (Infections and infestations) | 2 | 9 | 5
Decreased appetite (General disorders) | 1 | 4 | 7
Nasopharyngitis (Infections and infestations) | 1 | 1 | 8
Tachycardia (Cardiac disorders) | 0 | 2 | 7
Alanine aminotransferase increased (General disorders) | 1 | 7 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 2 | 4
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 0 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 4 | 1
Dry eye (Eye disorders) | 1 | 1 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 5 | 3
Vomiting (Gastrointestinal disorders) | 4 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Irritability (General disorders) | 1 | 2 | 1
Oedema peripheral (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 0
Pain (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1
Sluggishness (General disorders) | 0 | 1 | 0
Tenderness (General disorders) | 1 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 4
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 2
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Periumbilical abscess (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure increased (Investigations) | 2 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 0
Gamma-glutamyltransferase increase (Investigations) | 0 | 3 | 1
Heart rate increased (Investigations) | 0 | 1 | 1
Urinary sediment present (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 2 | 0
Weight increased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1
Heart sounds abnormal (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Salt craving (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 5 | 0
Migraine (Nervous system disorders) | 1 | 2 | 2
Sinus headache (Nervous system disorders) | 2 | 3 | 0
Somnolence (Nervous system disorders) | 3 | 1 | 1
Tremor (Nervous system disorders) | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 1
Sedation (Nervous system disorders) | 1 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 3 | 3
Abnormal dreams (Psychiatric disorders) | 0 | 2 | 0
Affect lability (Psychiatric disorders) | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 2
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Hostility (Psychiatric disorders) | 0 | 1 | 0
Illusion (Psychiatric disorders) | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 3 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Cystitis interstitial (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Hypomenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 2 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 3
Flushing (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No